CLINICAL TRIAL: NCT06343155
Title: Effect of Chronic Low Back Pain Treatment on Temporomandibular Disorder"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ikra Cakici, graduate student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-235
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Temporomandibular Disorder; Chronic Low-back Pain
Keywords: Temporomandibular disorder; Chronic low-back pain; Rocabado's exercise; Therapeutic lumbar exercise
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: There are two groups: Therapeutic group and Rocabado's group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercises (Experimental): Participants will be planned to participate in therapeutic lumbar exercises in groups of 5, in the morning and at noon, via the Zoom Platform in 40-minute sessions, 3 days a week, with a physiotherapist, for 6 weeks. Additionally, participants will do Rocabado's exercise at home. All exercises will be taught face to face in the first session. Online sessions with the physiotherapist will continue. A 5-minute warm-up and cool-down period and a 30-minute exercise period are planned. Patients will be asked to perform the exercises in 3 sets of 10-15 repetitions and will be allowed to rest for 10 seconds. Every exercise performed unilaterally will be performed bilaterally.
  Interventions: Other: Therapeutic Group; Other: Rocabado's Group
- Rocabado's Exercises (Active Comparator): Each exercise will consist of 6 sets and 6 repetitions.
  Interventions: Other: Rocabado's Group

INTERVENTIONS:
Other: Therapeutic Group — Pelvic tilt exercise:Participant will be supine position on the floor with your knees bent. Flatten your back against the floor by tightening your abdominal muscles and bending your pelvis up slightly. Lumbar flexion(single knee to chest): Participants will be supine position with knees bent and feet flat on the floor. The right knee will be brought closer to your chest and held with the hands. Lumbar flexion(double knee to chest) : Participants will be supine position with both legs flat on the floor. One hip and knee will be bent first to the chest, then the other to the chest. The knees will be grasped with the hands. Straight Leg Raise: Participants will be supine position with hips and legs comfortably on the floor. By contracting the quadriceps muscle the straight leg will be fixed. Inhaling slowly, the straight leg will be lifted six inches off the floor. Spine twist: Participants will turn their hips and knees to one side as much as possible in a supine position.
  Arms: Therapeutic Exercises
Other: Rocabado's Group — Rest position of tongue: Making a 'clucking' sound positions the tongue against the hard palate in the correct resting position for appropriate nasal and diaphragmatic breathing. Once the activity is practiced, the patient is to attempt to maintain appropriate tongue / jaw resting position throughout normal activity. Shoulder retraction:Sitting up nice and tall, squeeze your shoulder blades back and together. Stabilized head posture:Place your hands behind your hand with fingers interlocked.Gently bring head forward with gentle overpressure from hands.Axial extension of the neck: Sitting up nice and bring your chin backward as if trying to make a double chin. Rotation control of temporomandibular joint: Place tongue at the roof of your mouth just behind your front teeth and place fist underneath chin. Gently open mouth into fist and hold for a few seconds. Rhythmic stabilization:Patients apply resistance to opening, closing, and lateral deviation with the jaw in a resting position.

SUMMARY:
According to the information obtained from clinical studies, it has been stated that Temporomandibular Disorder (TMD) is associated with chronic low back pain (LBP). In this study, participants will be divided into two groups. Only Rocabado's exercise will be given to the Rocabado's group (RG), and Rocabado's and therapeutic lumbar exercises will be given to the therapeutic group (TG). Warm-up exercises will be given before starting the exercises with the therapeutic group, and cool-down exercises will be given after the exercises with the therapeutic group. At the end of the sixth week, the effect of therapeutic lumbar exercises on TMD pain and function will be evaluated.

DETAILED DESCRIPTION:
Studies indicate that TMD could coexist with low back pain. It has been proven in studies that physiotherapy reduces inflammation, joint pain, and mandibular movement limitation in TMD patients. The most common exercise known for TMD is defined as Rocabado's exercise 6x6. Each exercise is given in 6 sets of 6 repetitions. Rocabado's described techniques to facilitate neuromuscular stabilization using repeated lateral deviation movements. This technique can be used as a proprioceptive exercise method to increase functionality in areas where there is no pain. For patients with low back pain, our treatment goal is to minimize bed rest and restore functionality as soon as possible. Physiotherapy is recommended for patients with low back pain, and an exercise program is created according to the reasons and demands of the patients. There are many different intervention options, such as aerobic exercises, stretching exercises, and muscle building. Therapeutic exercises show positive results in low back and neck pain. In studies conducted in the treatment of TMD, the effect of therapeutic exercises on pain is still not fully known. Our aim in our study is to examine the effect of chronic low back pain treatment on temporomandibular disorder. Participants will be divided into two groups: the therapeutic group and the Rocabado's group. The therapeutic group will receive therapeutic lumbar exercises via remote online video for 6 weeks and will additionally be asked to do the Rocabado's exercise. Rocabado's exercises will be given to the Rocabado's group only as home exercises. In order to compare the effects of these techniques with each other, pre-treatment and post-treatment evaluations will be made for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 23-65
* Pain in the Temporomandibular Joint area for at least 3 months
* Participants had low back pain complaints for at least 6 months and were diagnosed with chronic low back pain.

Exclusion Criteria:

* History of trauma, anatomical deformities and fractures,
* Diagnosed orthopedic or rheumatological diseases,
* Acute trauma or infection in relevant areas,
* Pregnancy,
* Having received TMD treatment or been included in a physiotherapy program in the last 6 months,
* History of vertebral fracture in the last 6 months,
* Individuals with a history of surgery in the lumbar region.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-11 (Estimated); Primary Completion 2024-05-27 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Temporomandibular Joint Range of Motion Measurement (ROM) | six week
  Pain-free Mouth Opening (PMO):A premeasured mm caliper was attached to each participant's chin as a reference. Each participant will be instructed to open their mouth as wide as possible to the point where there is no pain.Maximum Unassisted Mouth Opening(MAO) It will be defined as the maximum distance a subject can open his mouth without feeling any pain. After the patient opens his mouth wide in this way, mouth opening will be measured.Maximum Assisted Mouth Opening(MAO): Once the patient is this open, the investigator will place his or her fingers on the patient's upper and lower central incisors, forcing the patient's mouth to open wider. Right Lateral Movement (RML)-Left Lateral Movement (LLM): Lateral right and left movements:Lateral right and left movements: For these measurements it is recommended the demarcation of two reference points, on the maxilla and mandible, close to the midline

SECONDARY OUTCOMES:
The Jaw Functional Limitation Scale 20 (JFLS-20) | six week
  The Jaw Functional Limitation Scale 20 (JFLS-20) will be used to measure changes in functional disability. The JFLS has 3 subcomponents: mastication, vertical jaw mobility, and emotional and verbal expression. The Jaw Functional Limitation Scale 20 (JFLS20) has a score range of 1 to 200, with higher scores indicating worsening jaw function.
Oral Health Impact Profile - 14 (OHIP-14) | six week
  Quality of life was measured using 14 item OHIP-14 comprising 7 different domains (functional limitation, physical pain, psychological discomfort, psychological disability, physical disability, social disability, and handicap) [10]. Each domain was assessed by two questions, scored using a 5-point Likert scale (0 = never to 4 = very often). The total OHIP-14 score was derived by a summing of the domain scores. A higher score indicates a poorer quality of life

OTHER OUTCOMES:
The short-form McGill Pain Questionnaire (SF-MPQ) | six weeks
  The short-form McGill Pain Questionnaire (SF-MPQ). Descriptors 1-11 represent the sensory dimension of pain experience and 12-15 represent the affective dimension. Each descriptor is ranked on an intensity scale of 0=none, 1=mild, 2=moderate, 3=severe. The Present Pain Intensity of the standard long -form McGill Pain Questionnaire and the visual analogue are also included to provide overall intensity scores.
Graded Chronic Pain Scale 2.0 total (GCPS 2.0) | six week
  GCPS 2.0 is a multidimensional measurement instrument that can provide information about the persistence of pain while determining both pain intensity and disability level. The scale asks about pain intensity for a period of the last 6 months. To measure the persistence of pain, the first item was added, which asks about the pain days experienced in the last 6 months. Other items ask about the situation in the one months period. In the converted form, there are 8 items. Items 2, 3, 4 measure pain intensity and items 5, 6, 7, 8 measure disability level.
Visual Analog Scale | six week
  The Visual Analogue Scale (VAS) will be measured low back pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark.

CONTACTS AND LOCATIONS:
Overall Officials: İkra Çakıcı, MD, Principal Investigator — Medipol University; Gizem Ergezen Şahin, Asst. Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Cakici I, Sahin GE. Exercise based multisite pain management in temporomandibular dysfunction and chronic low back pain: a randomized controlled trial. Physiother Theory Pract. 2025 Oct;41(10):2191-2201. doi: 10.1080/09593985.2025.2507848. Epub 2025 May 25. PMID 40415287